CLINICAL TRIAL: NCT07018453
Title: A Randomized, Open-label, Treat-to-target, Parallel-Controlled Phase II Clinical Study Investigating the Efficacy and Safety of SHR-3167 and Insulin Degludec in Type 2 Diabetic Subjects Treated With Basal Insulin With or Without Oral Antidiabetic Drugs
Brief Title: A Study Comparing SHR-3167 and Insulin Degludec in Type 2 Diabetic Subjects Treated With Basal Insulin With or Without Oral Antidiabetic Drugs
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3167-202
Record Dates: First submitted 2025-06-05; First posted 2025-06-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-3167 Group A (Experimental)
  Interventions: Drug: SHR-3167
- SHR-3167 Group B (Experimental)
  Interventions: Drug: SHR-3167
- Insulin Degludec Group (Active Comparator)
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: SHR-3167 — SHR-3167 Injection.
  Arms: SHR-3167 Group A; SHR-3167 Group B
Drug: Insulin Degludec — Insulin Degludec Injection.
  Arms: Insulin Degludec Group

SUMMARY:
The purpose of this study is to evaluate the glycemic control and safety of SHR-3167 and Insulin Degludec in type 2 diabetic participants treated with basal insulin with or without oral antidiabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 - 65 years old at the time of signing informed consent.
2. Diagnosed with type 2 diabetes mellitus (T2DM) for at least 6 months prior to the day of screening.
3. Treatment with basal insulin with or without oral antidiabetic drugs at least 90 days prior to the day of screening.
4. 6.5% ≤ HbA1c ≤ 10.0% at screening.

Exclusion Criteria:

1. Uncontrollable hypertension (with or without antihypertensive treatment) : systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg at screening.
2. Diagnosed or suspected with type 1 diabetes mellitus, latent autoimmune diabetes mellitus in adult (LADA), other special types of diabetes or secondary diabetes.
3. Known or suspected allergy or intolerance to the test drug or excipient.
4. There was a history of diabetic ketoacidosis or hyperglycemic hyperosmolar state within the previous 6 months.
5. There is acute or chronic hepatitis, liver cirrhosis, or a history of other serious liver diseases other than non-alcoholic fatty liver disease.
6. There is hyperthyroidism or hypothyroidism requiring treatment.
7. Malignancy within 5 years prior to screening or high risk of recurrence.
8. Those who have a history of severe cardiovascular and cerebrovascular diseases within 6 months before screening.
9. Participated in clinical trials of any drug or medical device within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) from baseline. | 16 weeks.

SECONDARY OUTCOMES:
Proportion of subjects with glycosylated hemoglobin (HbA1c) < 7.0% from baseline. | 16 weeks.
Change in fasting plasma glucose (FPG) from baseline. | 16 weeks.
Change in self-measured (capillary) blood glucose (SMBG) from baseline. | 16 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided